CLINICAL TRIAL: NCT06901778
Title: Adaptive Behavioral Intervention Application for Weight Control in Obese/Overweight Endometrial Cancer Patients in Fertility Preservation:A Randomized Clinical Trial
Brief Title: Application-Assisted Weight Management in Endometrial Cancer Fertility Preservation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaodan Li, associate professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB550-001
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer; Mobile Applications; Weight Management
Keywords: Endometrial Neoplasms; Mobile Applications; Weight Loss
MeSH Terms: conditions — Endometrial Neoplasms; Weight Loss | interventions — Amyloid Precursor Protein Secretases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): ① Implementation of the DEAR weight management model; ② Comprehensive coverage of the intelligent APP on the user end, and reinforcement of the regular interactive feedback and supervision mechanism of the medical team through the APP; ③ Provision of routine post-discharge care plans and follow-up programs.
  Interventions: Behavioral: DEAR weight management; Behavioral: Standardized discharge care plan and follow-up schedule; Behavioral: Implementation of the weight management mobile health application + Enhance the regular interaction, feedback, and supervision mechanism between medical teams and apps
- Control Group (Other): ① Implementation of the DEAR weight management model; ② Participants autonomously select functional modules of the weight management APP based on individualized health needs; ③ Provision of routine post-discharge care plans and follow-up programs.
  Interventions: Behavioral: DEAR weight management; Behavioral: Standardized discharge care plan and follow-up schedule; Behavioral: Implementation of the weight management mobile health application

INTERVENTIONS:
Behavioral: DEAR weight management — In the DEAR weight management model:
  D (Diet) refers to dietary management, primarily based on a calorie-restricted balanced diet; E (Exercise) refers to exercise management, guided by the 10th edition of the ACSM Exercise Testing and Prescription Guidelines and the 2017 National Fitness Guidelines. Exercise prescriptions are tailored to the patient's daily activity levels (light, moderate, and vigorous) to match the corresponding intensity levels; A (Accompany) refers to peer education, which involves using peer education methods to provide health education for patients, build confidence, and alleviate anxiety; R (Refresh) refers to rejuvenation, which involves correcting unhealthy dietary and exercise habits and establishing good lifestyle practices.
Behavioral: Standardized discharge care plan and follow-up schedule — Standardized discharge care plan and follow-up schedule providing patients and their families with professional and feasible pre-discharge education on disease-related knowledge, dietary and exercise recommendations, daily living advice, and psychological support to help patients establish healthy behaviors. Patients are provided with printed health education materials and a handbook on health and disease knowledge. A WeChat communication group is established to promptly answer patients' questions, encourage peer-to-peer experience sharing, and conduct regular telephone follow-ups and questionnaire surveys after discharge.
Behavioral: Implementation of the weight management mobile health application — Patients undergoing weight management are instructed to download the app from the app store (compatible with both iOS and Android platforms). Users in the control group can independently register and log in using their mobile phone numbers to access and use the app. The app will create an electronic health record for weight management for each user. Users can input their weight-related information, and the app features a data analysis function that displays weight trends through charts (e.g., BMI calculation and personal weight change curves). The app interface also provides professional guidance on diet and exercise, such as food calorie information, customized nutritional meal plans, and specialized exercise programs with training courses. By offering educational articles and instructional videos, the app aims to promote correct weight management concepts, disseminate scientific health knowledge, and enhance self-efficacy in weight loss.
  Arms: Control Group
Behavioral: Implementation of the weight management mobile health application + Enhance the regular interaction, feedback, and supervision mechanism between medical teams and apps — Based on the intelligent app's comprehensive coverage on the user side and integrating the ABI concept, the app dynamically adjusts intervention strategies. This is achieved by real-time collection and analysis of user behavior data, providing users with all around and personalized weight management support across diet, exercise, psychological support, etc., thereby enhancing the effectiveness and sustainability of interventions. The research team has formed a professional and experienced medical team. All members hold a bachelor's degree or above and possess rich clinical weight management experience. Through the app, they provide users with scientific and rigorous supervision and guidance. During weight loss, users can obtain accurate, professional answers and personalized adjustment advice in real-time via the app's question-asking column if they encounter any problems.
  Arms: Experimental Group

SUMMARY:
This study is a single-center, prospective, randomized controlled trial targeting endometrial cancer (EC) patients undergoing fertility-sparing treatment at Peking University People's Hospital from March 2025 to March 2027. The aim is to evaluate the efficacy of an intelligent mobile application (APP) based on the Adaptive Behavioral Intervention (ABI) framework in weight management for obese or overweight endometrial cancer patients receiving fertility preservation therapy. Additionally, the study seeks to explore its potential advantages in improving body mass index (BMI), tumor regression, and glucose and lipid metabolism profiles.

DETAILED DESCRIPTION:
Endometrial cancer is one of the most common malignancies of the female reproductive tract, with obesity being a closely associated factor in its development and progression. According to the American Cancer Society, 57% of endometrial cancer cases are linked to obesity, and a 5-unit increase in body mass index (BMI) elevates the risk of EC by 50%. Overweight or obesity adversely impacts treatment efficacy and reduces survival rates in EC patients. In recent years, the incidence of EC has shown a trend toward younger populations, posing significant threats to the health and quality of life of patients undergoing fertility-sparing treatment. The Adaptive Behavioral Intervention (ABI) framework emphasizes real-time adjustments based on individual feedback and progress to optimize behavioral change and health outcomes. Integrating smart application (APP) technology can provide more convenient and personalized weight management support for EC patients undergoing fertility preservation. By continuously collecting and analyzing behavioral data, the intervention strategy can be dynamically tailored, thereby enhancing the effectiveness and sustainability of the intervention. Currently, there is a paucity of research on comprehensive weight management interventions incorporating intelligent APPs for obese or overweight EC patients in fertility-sparing treatment. This study aims to investigate the efficacy of an ABI-based smart APP in weight management for this population through a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 kg/m²
* Histologically confirmed endometrial carcinoma via diagnostic curettage, hysteroscopic endometrial biopsy, or needle biopsy
* Clinical FIGO 2009 stage IA disease: No evidence of extrauterine metastasis or myometrial invasion on imaging (MRI/CT)
* ECOG < 2
* Active desire to preserve fertility
* Fertility-preserving treatment
* Willingness to participate and signed informed consent

Exclusion Criteria:

* High-grade or p53-mutated (p53mut) endometrial cancer
* Currently using weight-loss medications
* Pregnant or breastfeeding
* Presence of communication barriers that prevent understanding and participation in the informed consent process
* Participation in other weight-loss programs
* Inability to safely engage in unsupervised physical activities
* Undergoing anticoagulant therapy that may affect body composition, weight, or energy expenditure
* Severe comorbidities: urinary system stones, history of renal failure or severe renal insufficiency, familial dyslipidemia, severe liver disease, chronic metabolic acidosis, history of pancreatitis, severe diabetes, active gallbladder disease, fat malabsorption, severe cardiovascular and cerebrovascular diseases
* Presence of unstable medical conditions: uncontrolled hypertension, diabetes, unstable angina, transient ischemic attack, other cancers currently under treatment, Crohn's disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  Use the Inbody720 to measure height and weight and calculate BMI according to the formula "BMI (= weight (kg)/height² (m²)"

SECONDARY OUTCOMES:
Waist circumference (WC) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  Physiological parameter measured with the subject's body upright, abdomen relaxed, both arms hanging down naturally, feet together, and the tape measure placed around the waist; the height was adjusted to the horizontal plane passing through the midpoint of the line between the lower edge of the rib arch and the iliac crest in the mid-axillary line
Hip circumference (HC) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  Measured with the subject's body upright, taking the circumference of the body at the horizontal position of the uppermost point of the hip
Waist-to-height ratio (WHtR) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  Calculate WHtR according to the formula "WHtR= waist circumference (cm)/height (cm)= waist circumference (cm)/height (cm)"
Waist-to-hip ratio (WHR) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  Calculate WHR according to the formula "WHR=waist circumference (cm)/hip circumference (cm)"
Body shape index (ABSI) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  Calculate ABSI according to the formula "ABSI= (waist)/([BMI]^2/3×height^1/2)"
Body roundness index (BRI) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  Calculate BRI according to the formula "BRI= waist/BMI"
Visceral fat index (VAI) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  Calculate VAI according to the formula "VAI= waist/(36.58 + 1.89 × BMI) × triglyceride (TG) level/0.81 × 1.52/high density lipoprotein (HDL) level"
Lipid accumulation index (LAP) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  Calculate LAP according to the formula "LAP= = (waist circumference - 58) × TG level"
Triglycerides | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Cholesterol | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
High density lipoprotein (HDL) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Low density lipoprotein (LDL) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Fasting glucose | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Fasting insulin (FINS) | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Glycated hemoglobin | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Weight efficacy | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  The Weight Efficacy Lifestyle Questionnaire-Short Form (WEL-SF) was utilized to assess Weight Efficacy. This validated instrument comprises 8 items, scored on a scale of 0 to 80, with higher scores indicating greater self-efficacy in weight management
Exercise adherence | Baseline / Month 3 of intervention / Month 6 of intervention / Month 9 of intervention / Month 12 of intervention
  The Chinese-translated version of the Exercise Adherence Rating Scale (EARS) was employed to evaluate Exercise Adherence. The EARS consists of 16 items, scored from 0 to 64, with higher scores reflecting stronger exercise adherence. Items 1, 3, 5, 9, 13, 14, and 16 are reverse-scored to ensure psychometric accuracy
Complete response (CR) | One year of intervention
  Complete remission indicated by complete endometrial regression and interstitial metaplasia-like changes on histopathology after treatment (without any endometrial atypical hyperplasia or endometrioid adenocarcinoma lesions, as clarified by pathologists)
Application usage frequency | one year of intervention
  The backend retrieves user application usage days data within a year, defining application usage frequency by the number of application usage days.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodan Li, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China